CLINICAL TRIAL: NCT03507998
Title: A Phase 1 Open-label Dose Escalation Study of CGX1321 in Subjects With Advanced Gastrointestinal Tumors
Brief Title: Phase 1 Dose Escalation Study of CGX1321 in Subjects With Advanced Gastrointestinal Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Curegenix Inc. (Industry)
Collaborators: Guangzhou Curegenix Co. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGX1321-102
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Adenocarcinoma; Gastric Adenocarcinoma; Pancreatic Adenocarcinoma; Bile Duct Carcinoma; Hepatocellular Carcinoma; Esophageal Carcinoma; Gastrointestinal Cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Carcinoma, Hepatocellular; Esophageal Neoplasms; Gastrointestinal Neoplasms | interventions — CGX1321

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CGX1321 Dosing (Experimental): Dose Escalation Phase: Ascending doses of CGX1321 will be administered by cohort to determine the maximum tolerated dose. Patients will receive CGX1321, once daily, orally, for 3 weeks (21 days) followed by a one week (7 day) washout period in each 28 day cycle, according to the cohort they are assigned.
  Dose Expansion Phase: Patients will receive the recommended dose (identified in the Dose Expansion Phase) of CGX1321
  Interventions: Drug: CGX1321

INTERVENTIONS:
Drug: CGX1321 — CGX1321 capsules for oral administration

SUMMARY:
This is a multi-center, open label, repeat dose, Phase 1 study consisting of a Dose Escalation Phase and a Dose Expansion Phase to evaluate safety, pharmacokinetics, and clinical activity.

DETAILED DESCRIPTION:
The purpose of the Dose Escalation Phase is to examine the safety and determine the maximum tolerated dose of CGX1321 when administered to subjects with advanced GI tumors that have relapsed or are refractory to or not considered medically suitable to receive standard of care treatment.

Once the dose is identified in the Dose Escalation Phase, the Dose Expansion Phase will start. The purpose of the Dose Expansion Phase is to continue to examine the safety and confirm the final Phase 2 dose of CGX1321 when administered to subjects with advanced GI tumors who meet the entry criteria.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-diagnosed advanced Gl tumors, such as colorectal adenocarcinoma, gastric adenocarcinoma, pancreatic adenocarcinoma, bile duct carcinoma, hepatocellular carcinoma, esophageal carcinoma that have relapsed or are refractory to or are not considered medically suitable to receive standard of care treatment
* Eastern Cooperative Oncology Group (ECOG) score of 0 - 1
* Minimum estimated life expectancy of 3 months
* Adequate organ function
* Recovery from prior treatment-related toxicities
* Ability to swallow capsules
* Willingness for subjects of reproductive potential to use adequate methods of contraception during and for 3 months after study treatment

Exclusion Criteria:

* Prior exposure to a WNT inhibitor
* Received previous therapy for malignancy within 21 days
* Major surgery within 4 weeks of first dose of study drug
* Radiotherapy within 2 weeks of first dose of study drug
* Significant GI or variceal bleeding or subdural hematoma within 3 months of treatment start
* Uncontrolled central nervous system metastases or leptomeningeal metastases
* Requirement for immunosuppressive agents (must be off for at least 7 days)
* Currently receiving medications that are known CYP3A4/5 inhibitors. Patients currently receiving medications of known inducers of CYP3A4/5 or substrates of CYP2C8/9 and CYP1A2 may be excluded.
* Bone abnormalities
* Hypercalcemia
* Cardiac abnormalities
* Known human immunodeficiency virus positive, or active hepatitis A, B or C
* History of additional prior malignancy with the exception of surgically cured carcinomas such as skin, prostate, bladder, thyroid, cervix or other carcinomas in situ
* Active systemic infection requiring intravenous antibiotics within 2 weeks of treatment start
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2017-06-17 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events and/or abnormal laboratory values that are related to treatment | 21 months

SECONDARY OUTCOMES:
CGX1321 maximum or peak concentration | 30 days
CGX1321 minimum or trough concentration | 30 days
CGX1321 time to maximum concentration | 30 days
CGX1321 half life | 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: No